CLINICAL TRIAL: NCT05850780
Title: Clinical and Radiographic Evaluation of Laser Photobiomodulation Pulpotomy of Primary Molars in Children (A Randomized Controlled Clinical Trial)
Brief Title: Clinical and Radiographic Evaluation of Laser Photobiomodulation Pulpotomy of Primary Molars in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aliaa Hamouda (Other)
Responsible Party: Sponsor-Investigator, Aliaa Hamouda, Assistant Lecturer of Pediatric Dentistry, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #12
Record Dates: First submitted 2023-04-29; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Pulpitis; Pulpotomy
MeSH Terms: conditions — Pulpitis | interventions — Low-Level Light Therapy; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation (Experimental)
  Interventions: Device: Photobiomodulation
- Mineral Trioxide Aggregate (MTA) (Active Comparator)
  Interventions: Drug: MTA

INTERVENTIONS:
Device: Photobiomodulation — A diode laser (Sirolaser blue laser system, Sirona Dental Systems GmbH, Fabrikstraße 31, 64625 Bensheim, Germany) Wavelength 660 nm will be used, and the laser parameters will be set as follows: Power 0.1 W, energy 6 J, Continuous wave; energy Tip area 0.5 cm2, fluence 12 J/cm2 will be applied to the surface of the pulp stumps for 60 seconds. The pulp chamber will then be filled with reinforced zinc oxide-eugenol (IRM, Dentsply, Mount Waverley, Australia) to ensure proper sealing.
  Then, each tooth in both groups will finally be restored with a stainless-steel crown (SSC)40 (3M/ESPE, St. Paul, Minn., USA) in the same visit, which will be cemented onto the tooth using glass ionomer cement.
  Finally, reapplication of laser with the same parameters will be done around inserted crowns to promote tissue healing and decrease post operative pain.
  Arms: Photobiomodulation
Drug: MTA — Three parts of MTA powder will be mixed with one part of distilled water to obtain paste. This mixture will then be placed on the radicular pulp stumps and condensed lightly with a moistened cotton pellet. then the access cavities will be sealed with glass ionomer cement
  Arms: Mineral Trioxide Aggregate (MTA)

SUMMARY:
This study aimed to evaluate the clinical and radiographic outcomes of photobiomodulation pulpotomy compared to MTA pulpotomy in primary molars in children.

ELIGIBILITY:
Inclusion Criteria:

* Children with dental behavior score of 3 or 4 according to the Frankel behavior rating scale.
* Patients whom their maxillary primary molars are indicated for pulpotomy and SSC restoration.
* Lack of history of allergy to the materials used for anesthesia and sulfite.
* Children free of any systemic disease or special health care needs (ASA 1).
* Completion of the written informed consent form by parents/guardian.

Exclusion Criteria:

* Children who receive any analgesic drugs at least 24 hours before treatment.
* Any inflammation or lesion in the injection site
* Patients who have previous bad experience of dentistry were excluded to eliminate the possible impact of the child's previous painful or stressful experiences
* Child coming for emergency treatment of pain.
* If hemostasis is not achieved within five minutes after application of moist cotton pellet directly to the pulp stumps
* If radicular pulp tissue was not vital due to the presence of suppuration or purulent necrosis (pus discharge).

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Clinical success of pulpotomy | up to 12 months
  Patients will be assessed and the presence of any adverse clinical signs or symptoms pain, or swelling will be considered clinical criteria of failure
Radiographic success of pulpotomy | up to 12 months
  Periapical x-ray will be performed and the presence of any any periapical radiolucency, furcation involvement, widening of periodontal ligament space (PDL), and pathologic internal/external root resorption will be considered radiographic failure.
Tissue healing | 24 hours
  Tissue healing after stainless steel crown (SSC) insertion will be assessed according to gingival index scale to determine the gingival condition around the inserted SSC. The adopted Löe and Silness gingival index scale ranges from 0 to 3 for the buccal, lingual, mesial and distal surfaces, and will be scored as follows: 0 indicates no inflammation and healthy gums; 1 indicates mild inflammation where there is slight color changes, slight edema and no bleeding on probing; 2 indicates moderate inflammation where there is edema with slight redness and bleeding upon probing; and 3 indicates severe inflammation where there is severe edema, redness, presence of ulceration and a tendency for spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Hamouda, MSc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Amani Khalil, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Laila El-Habashy, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt